CLINICAL TRIAL: NCT06930677
Title: A Prospective, Single-arm, Multinational, Multi-center, Clinical Study to Evaluate the Performance and Safety of Musculoskeletal Embolization Using NBGM200 in Patients With Knee Degenerative Osteoarthritis
Brief Title: Study in Patients With Knee Osteoarthritis Treated by Embolization Using NBGM200
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Next Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAME 003; GENTILLE (Other: Elisabeth-Tweesteden Hospital)
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthritis (Knee OA)
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSK embolization (Experimental)
  Interventions: Device: embolization therapy

INTERVENTIONS:
Device: embolization therapy — MSK embolization

SUMMARY:
Study in patients with knee osteoarthritis treated by embolization using NBGM200

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis proven by MR-imaging

Exclusion Criteria:

* Current local infection
* Life expectancy less than 6 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome score (KOOS-12) | 6 months post treatment
  Knee Injury and Osteoarthritis Outcome score (KOOS-12) is to evaluate the pain, function and quality of life. The total score ranges from 0 to 100, where higher scores indicate better outcomes.

SECONDARY OUTCOMES:
Visual Analog Scale(VAS) | 6 months post treatment
  Visual Analog Scale(VAS) is to evaluate the pain from 0 to 10. Higher scores indicate worse outcomes, representing more severe pain
Whole Organ Magnetic Resonance Imaging Score (WORMS) | 6 months post treatment
  Whole Organ Magnetic Resonance Imaging Score (WORMS) is a semi-quantitative scoring method for multi-feature, whole-organ evaluation of knee OA based on MRI. The total score ranges from 0 to 332, with higher scores indicating worse outcomes.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (2):
  - University Hospital Ghent, Ghent
  - Uz Leuven, Leuven
- Elisabeth-Tweesteden Hospital, Tilburg, Netherlands